CLINICAL TRIAL: NCT02947334
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled, Parallel-group Study To Assess The Efficacy, Safety And Tolerability Of Bococizumab (Pf-04950615) In Asian Subjects With Primary Hyperlipidemia Or Mixed Dyslipidemia At Risk Of Cardiovascular Events
Brief Title: Efficacy And Safety Of Bococizumab For Lipid Lowering In Asian Hypercholesterolemia Subjects
Acronym: SPIRE-ASIA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1481047
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Primary Hyperlipidemia or Mixed Dyslipidemia
MeSH Terms: interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bococizumab (Experimental): Bococizumab Q2wks
  Interventions: Biological: Bococizumab
- Placebo (Placebo Comparator): Bococizumab placebo Q2wks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Bococizumab — Bococizumab PFS
  Other Names: RN316
  Arms: Bococizumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a Phase 3, double blind, placebo controlled, randomized, stratified, parallel group, multi-center clinical trial designed to compare the efficacy and safety of bococizumab 150 mg SC Q2wks to placebo for LDL-C lowering in subjects with primary hyperlipidemia or mixed dyslipidemia at high or very high risk for CV events. The study will enroll a total of approximately 750 subjects from 4 - 5 Asian countries/areas (including China mainland); of which approximately 600 subjects will be from sites in China. Subjects will be randomized into a bococizumab treatment arm and a placebo arm in a 1:1 ratio.

DETAILED DESCRIPTION:
After providing consent, subjects will enter a screening period of approximately 28 days to verify eligibility for the trial. Eligible subjects will be considered enrolled and progress to the Randomization visit. Results from screening evaluations will be reviewed and only subjects who continue to meet all eligibility criteria will be randomized. Randomized subjects will enter the 12-week treatment period, followed by a 40-week long-term treatment period and a 6 week follow-up, for a total of 58 weeks (approximately 14 months) study participation. Subjects will attend clinic visits as shown in the Schedule of Activities. Subjects will be randomized to receive either 150 mg Q2wks of bococizumab or placebo in a 1:1 ratio. Lipid levels will be blinded to the investigator and staff, subject and sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at the age or over 18 years of age.
* With primary hyperlipidemia or mixed dyslipidemia.
* Treated with stable daily dose of statins
* At high or very high risk of incurring a CV event
* Fasting LDL-C >=70 mg/dL (1.81 mmol/L) for subjects on the highest approved dose of statins; Fasting LDL C >=77 mg/dL (1.99 mmol/L) for subjects not on highest approved dose.
* Fasting TG ≤400 mg/dL (4.51 mmol/L)

Exclusion Criteria:

* Prior exposure to bococizumab or other investigational PCSK9 inhibitor
* NYHA class IV, or Left Ventricular Ejection Fraction <25%
* Poorly controlled hypertension
* History of hemorrhagic stroke or lacunar infarction resulting in a stroke
* Untreated hyperthyroidism or TSH >1 × ULN
* Undergoing apheresis or have planned start of apheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-31 (Estimated); Primary Completion 2019-05-03 (Estimated); Study Completion 2019-05-03 (Estimated)

PRIMARY OUTCOMES:
• Percent change from baseline in fasting LDL-C | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481047&StudyName=A%20Phase%203%20Double-blind%2C%20Randomized%2C%20Placebo-controlled%2C%20Parallel-group%20Study%20To%20Assess%20The%20Efficacy%2C%20Safety%20And%20Tolerability%20Of%20Bococizumab%20%28pf-04950615%29%20In%20Asian%20Subjects%20With%20Primary%20Hyperlipidemia%20Or%20Mixed%20Dyslipidemia%20At%20Risk%20Of%20Cardiovascular%20Events
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481047&StudyName=A+Phase+3+Double-blind%2C+Randomized%2C+Placebo-controlled%2C+Parallel-group+Study+To+Assess+The+Efficacy%2C+Safety+And+Tolerability+Of+Bococizumab+%28pf-04950615%29+In+Asian+Subjects+With+Primary+Hyperlipidemia+Or+Mixed+Dyslipidemia+At+Risk+Of+Cardiovascular+Events